CLINICAL TRIAL: NCT02090283
Title: An Open Label Extension, Multi-Center, Study to Evaluate the Safety of SD-101 Cream in Subjects With Epidermolysis Bullosa
Brief Title: Open-Label Extension Study to Evaluate the Safety of SD-101 Cream in Participants With Epidermolysis Bullosa
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor voluntarily recalled SD-101 and terminated the study due to GMP deficiencies identified during an FDA inspection at the site of the manufacturer.
Sponsor: Scioderm, Inc. (Industry)
Collaborators: Amicus Therapeutics (Industry); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-004; 1R01FD005093-01 (FDA)
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Epidermolysis Bullosa
Keywords: Amicus Therapeutics; Scioderm, Inc.; Recessive Dystrophic; Junctional non-Herlitz; Epidermolysis Bullosa; Simplex; SD-101 6%; SD-101-6.0; Allantoin 6%; Zorblisa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD-101 Dermal Cream (6%) (Experimental): All participants applied SD-101 dermal cream topically, once a day, to the entire body for the duration of the study.
  Interventions: Drug: SD-101 dermal cream (6%)

INTERVENTIONS:
Drug: SD-101 dermal cream (6%) — SD-101 is a white, crystalline powder that is formulated within an odorless, soft, white cream base. SD-101-6.0 cream contains allantoin, a diureide glyoxylic acid, at a concentration of 6% and other excipients.
  Other Names: SD-101; SD-101-6.0; Zorblisa

SUMMARY:
The purpose of this study was to assess the continued safety of topical use of SD-101 cream (6%) in participants with Epidermolysis Bullosa (EB).

Funding Source: FDA Office of Orphan Products Development

DETAILED DESCRIPTION:
This was an open-label extension study to assess the continued safety of topically applied SD-101 dermal cream (6%) in participants with Simplex, Recessive Dystrophic, and Junctional non-Herlitz EB.

SD-101 dermal cream (6%) was applied topically, once a day to the entire body for the duration of the study. Participants who successfully completed the entire SD-003 study (NCT02014376) had the option to roll over into the SD-004 study (NCT02090283). The baseline visit occurred at the final visit date for the SD-003 study. The body surface area (BSA) coverage of blisters and lesions assessment made at the final SD-003 study visit were used as the baseline information at the baseline visit for the SD-004 study. Participants returned to the study site for the following 13 visits (36 months) to have BSA assessed. BSA was assessed at all subsequent scheduled study center visits. Scheduled study center visits occurred every 6 months after Month 36 (Month 42, 48, and so on). After completion of Month 36, the next participant visit (Month 39) was a phone call from the site to the participant. Telephone visits occurred every 6 months thereafter (Month 45, 51, and so on) and included assessment of adverse events and concomitant medications only. For female participants of childbearing potential, a urine pregnancy test was performed at Month 6 and every 6 months up to and including the final study visit.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the participant or participant's legal representative; if the participant is under the age of 18 but capable of providing assent, signed assent from the participant.
* Participant (or caretaker) must be willing to comply with all protocol requirements.
* Participant must have successfully completed the SD-003 study.

Exclusion Criteria:

* Participants who do not meet the inclusion criteria.
* Pregnancy or breastfeeding during the study. A urine pregnancy test will be performed at the final visit for SD-003 for female participants of childbearing potential.
* Females of childbearing potential who are not abstinent and not practicing a medically acceptable method of contraception.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Amicus Therapeutics
Locations (7):
- United States (7):
  - Palo Alto, California
  - Chicago, Illinois
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Chapel Hill, North Carolina
  - San Antonio, Texas
  - Seattle, Washington

REFERENCES:
- [Result] Paller A., Browning J., Aslam R., et al. Efficacy and Safety Results From a 24-Month, Open-Label Extension of a Phase 2b Dose-Ranging Study of SD-101 Cream in Patients With Epidermolysis Bullosa. Abstract presented at European Academy of Dermatology and Venereology, 26th Congress, Geneva, Switzerland, September 13-17, 2017.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 participants with epidermolysis bullosa (EB) were enrolled in this open-label, multi-center extension study. All enrolled participants had previously completed Study SD-003 (NCT02014376).
Pre-assignment Details: Analysis groups were defined based on prior treatment in Study SD-003: those who received placebo were allocated to the 'Placebo to SD-101-6.0' group, those who received SD-101-3.0 were allocated to the 'SD-101-3.0 to SD-101-6.0' group, and those who received SD-101-6.0 were allocated to the 'SD-101-6.0 to SD-101-6.0' group.
Groups:
- Placebo to SD-101-6.0: Participants who received placebo in Study SD-003 received SD-101-6.0 in this open-label extension study. SD-101-6.0 was applied topically, once a day, to the entire body.
- SD-101-3.0 to SD-101-6.0: Participants who received SD-101-3.0 in Study SD-003 received SD-101-6.0 in this open-label extension study. SD-101-6.0 was applied topically, once a day, to the entire body.
- SD-101-6.0 to SD-101-6.0: Participants who received SD-101-6.0 in Study SD-003 continued to receive SD-101-6.0 in this open-label extension study. SD-101-6.0 was applied topically, once a day, to the entire body.
Period: Overall Study
Arm/Group | Placebo to SD-101-6.0 | SD-101-3.0 to SD-101-6.0 | SD-101-6.0 to SD-101-6.0
Started | 17 | 15 | 10
Received At Least 1 Dose Of Study Drug | 17 | 15 | 10
Completed | 0 | 0 | 0
Not Completed | 17 | 15 | 10
Not completed — Withdrawal by Subject | 6 | 6 | 6
Not completed — Sponsor Terminated Study | 6 | 6 | 1
Not completed — Lost to Follow-up | 2 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Protocol Violation | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety: All participants who successfully rolled over into the SD-004 study from the SD-003 study and applied/were administered at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to SD-101-6.0 | SD-101-3.0 to SD-101-6.0 | SD-101-6.0 to SD-101-6.0 | Total
Number analyzed (Participants) | 17 | 15 | 10 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.29 (10.385) | 15.70 (15.928) | 8.10 (4.795) | 12.11 (11.945)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 18
  Male | 12 | 7 | 5 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 3 | 14
  Not Hispanic or Latino | 12 | 9 | 7 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 16 | 15 | 7 | 38
  Race: Black or African-American | 1 | 0 | 2 | 3
  Race: Asian | 0 | 0 | 1 | 1
EB Subtype [Count of Participants; unit: Participants]
  Simplex | 4 | 4 | 3 | 11
  Recessive Dystrophic | 10 | 8 | 6 | 24
  Junctional non-Herlitz | 3 | 3 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Treatment-emergent adverse events were defined as adverse events that started or worsened on or after baseline visit, which occurred at the final visit date for the SD-003 study. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From baseline to 30 days after last application of study drug (up to a maximum of 54 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo to SD-101-6.0 | SD-101-3.0 to SD-101-6.0 | SD-101-6.0 to SD-101-6.0
Number analyzed (Participants) | 17 | 15 | 10
Participants
  Any TEAE | 13 | 14 | 5
  Any TEAE Related to Study Drug | 1 | 1 | 0
  Any Fatal TEAE | 0 | 0 | 0
  Serious TEAE | 4 | 2 | 0
  Any TEAE Leading to Discontinuation | 1 | 1 | 0

2. Secondary Outcome: Change From Baseline In Body Surface Area Index (BSAI) Of Lesional Skin At Month 24
Description: Lesional skin was defined as areas that contained any of the following: blisters, erosions, ulcerations, scabbing, bullae, or eschars, as well as areas that were weeping, sloughing, oozing, crusted, or denuded. The percentage, ranging from 0% to 100%, of affected body surface area (BSA) was recorded for each defined body region (that is, head/neck, upper limbs, trunk [includes groin], and lower limbs), multiplied by the weighting factor, and then summed for all body regions to calculate the BSAI. The BSA for lesional skin was to be assessed by the same study physician on each visit for a particular participant. The mean change from baseline (final visit from the SD-003 study) in BSAI was assessed every 3 months. Only participants with data available for analysis at the specified time point are presented.
Time Frame: Baseline, Month 24
Population: Intent to Treat: All participants who successfully rolled over into the SD-004 study from the SD-003 study and applied/were administered at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of BSAI
Arm/Group | Placebo to SD-101-6.0 | SD-101-3.0 to SD-101-6.0 | SD-101-6.0 to SD-101-6.0
Number analyzed (Participants) | 9 | 9 | 3
percentage of BSAI | 1.99 (6.728) | -3.73 (6.152) | -9.50 (21.248)

ADVERSE EVENTS:
Time Frame: From baseline (Day 0) to 30 days after last application of study drug (up to a maximum of 54 months).
Arm/Group | Placebo to SD-101-6.0 | SD-101-3.0 to SD-101-6.0 | SD-101-6.0 to SD-101-6.0
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/17 | 2/15 | 0/10
Other Adverse Events (participants affected / at risk) | 13/17 | 13/15 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to SD-101-6.0 (N=17) | SD-101-3.0 to SD-101-6.0 (N=15) | SD-101-6.0 to SD-101-6.0 (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to SD-101-6.0 (N=17) | SD-101-3.0 to SD-101-6.0 (N=15) | SD-101-6.0 to SD-101-6.0 (N=10)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 2 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Myopia (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 0
Pain (General disorders) | 0 | 2 | 0
Application site pain (General disorders) | 0 | 1 | 0
Developmental delay (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 1 | 0
Skin infection (Infections and infestations) | 4 | 2 | 0
Ear infection (Infections and infestations) | 2 | 2 | 0
Influenza (Infections and infestations) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Wound infection (Infections and infestations) | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Bacterial disease carrier (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0
Stoma site cellulitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Pancreatic enzymes decreased (Investigations) | 1 | 0 | 0
Serum ferritin decreased (Investigations) | 1 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pseudosyndactyly (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Borderline personality disorder (Psychiatric disorders) | 0 | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0
Cyst removal (Surgical and medical procedures) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Results are presented for all participants who received SD-101 before the early termination of the study on 4 June 2018. The maximum study duration completed by at least 1 participant was 54 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT02090283/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT02090283/SAP_001.pdf